CLINICAL TRIAL: NCT05858801
Title: First Evaluation of a Craniofacial Peripheral Nerve Stimulation System in Chronic Migraine, an Early Feasibility Study
Brief Title: First Evaluation of a Craniofacial Peripheral Nerve Stimulation System in Chronic Migraine
Acronym: RELIEF
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Salvia BioElectronics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: SCI-02-CM
Record Dates: First submitted 2023-05-05; First posted 2023-05-15 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Chronic Migraine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PRIMUS (Experimental): PRIMUS system
  Interventions: Device: PRIMUS

INTERVENTIONS:
Device: PRIMUS — PRIMUS system

SUMMARY:
The purpose of this study is to demonstrate the safe use of the PRIMUS system in subjects with chronic migraine. This is a single-center, open label, prospective, early feasibility study to collect initial clinical data on the PRIMUS system for the treatment of chronic migraine.

ELIGIBILITY:
Main Inclusion Criteria:

* Able and willing to provide informed consent
* Age ≥ 18 years and ≤ 84 years at time of consent
* Documented Chronic Migraine, defined as at least eight migraine days/month, for at least 1 year.
* Developed migraine before the age of 50
* Documented failure of 3 or more other preventive therapies (failure meaning ineffective, provoked unacceptable side-effects or contra-indicated) from which at least 1 of the following 2: CGRP mAbs or Onabotulinumtoxin A
* Have at least 1 headache free day per month
* Stable on preventive migraine drugs and alternative treatment for at least three months prior to enrollment.
* Agree to refrain from starting new preventive migraine drugs or other preventive alternative migraine treatments, from 4 weeks before entering the baseline period throughout the duration of the study.
* MRI available (not older than 4 years prior to study enrollment) or willing to undergo an MRI to exclude structural lesions potentially causing headache
* Able and willing to complete a daily headache eDiary

Main Exclusion Criteria:

* Any other chronic primary or secondary headache disorder, unless they can clearly differentiate them from migraine attacks, based on the quality of pain and associated symptoms.
* Concomitant neuromodulation
* Previous failure to an implantable neuromodulation device for neurovascular headache
* Have an existing Active Implantable Medical Device nearby the implant location (e.g. DBS, cochlear implant, …)
* Metal implants in the skull (e.g. skull plates, seeds) nearby the implant.
* Have a pacemaker of implantable cardioverter defibrillator (ICD)
* Current Opioid Use, defined as one or more opioids on more than 4 days/month for 3 consecutive months.
* Use of botulinum toxin injections in the past 3 months.
* Women of childbearing age who are pregnant, nursing or not using contraception

Ages: 18 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2023-05-09 (Actual); Primary Completion 2023-12-09 (Actual); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Safety Evaluation | 30 days
  The primary safety assessment is the incidence of serious procedure- and/or device-related adverse events in all subjects at 30 days and at the end of the study.
  All adverse clinical events will be collected, coded, and reported, for the duration of the study according to the definitions of ISO 14155:2020.
Safety Evaluation | 12 months
  The primary safety assessment is the incidence of serious procedure- and/or device-related adverse events in all subjects at 30 days and at the end of the study.
  All adverse clinical events will be collected, coded, and reported, for the duration of the study according to the definitions of ISO 14155:2020.

CONTACTS AND LOCATIONS:
Locations (1):
- AZ Delta, Roeselare, Belgium

IPD SHARING:
Plan to Share IPD: No